CLINICAL TRIAL: NCT05099198
Title: Replication of the GRADE Diabetes Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-GRADE
Record Dates: First submitted 2021-06-25; First posted 2021-10-29 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sitagliptin: Reference group
  Interventions: Drug: Sitagliptin
- Glimepiride: Exposure group
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin dispensing claim is used as the reference
  Groups: Sitagliptin
Drug: Glimepiride — Glimepiride dispensing claim is used as the reference
  Groups: Glimepiride

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal than 30: days [0,0]
* Diagnosis of Type 2 Diabetes: days [- All Data, 0]
* 2+ recorded HbA1c levels: days [-365,0]
* Metformin use: days [-30, 0]

Exclusion Criteria:

* Type 1 or Secondary DM: days [-All Data, 0]
* Previous organ transplant: days [-All Data, 0]
* HIV/AIDS: days [-All Data, 0]
* History of bariatric surgery: days [-All Data, 0]
* Congestive heart failure: days [-All Data, 0]
* NYHA >=3: days [-All Data, 0]
* Pancreatitis: days [-All Data, 0]
* Medullary thyroid cancer/MEN-2: days [-All Data, 0]
* History of MI: days [-365, 0]
* Stroke: days [-365, 0]
* Coronary Revascularization: days [-365, 0]
* PTCA/Stenting/CABG: days [-365, 0]
* Trans myocardial revascularization: days [-365, 0]
* Carotid bypass: days [-365, 0]
* Cerebrovascular revascularization: days [-365, 0]
* PVD: days [-365, 0]
* CCI >=10: days [-365, 0]
* History of cancer, other than non-melanoma skin cancer: days [-1,825, 0]
* Treatment of metformin more than 10 years: days [-3,650, 0]
* Treatment with any diabetes drug other than metformin; PCOS; symptomatic hyperglycemia; pregnancy; gestational diabetes: days [-180, 0]
* History of hemolytic anemia; history of severe liver disease; current alcoholism; chronic transfusion requirement; ESRD: days [-180, 0]
* Oral, IV, or IM cortisone, hydrocortisone, prednisone, methylprednisone, or dexamethasone: days [-90, 0]
* Treatment with atypical antipsychotics, language barriers, nursing home, or missing age or gender: days {-180, 0]
* Hospitalization with length of stay >3 days: days [-30, 0]

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who have previously been treated with metformin.
Sampling Method: Non-Probability Sample
Enrollment: 6403 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Time until failure to maintain metabolic control | Through censoring or study completion, up to 765 days after cohort entry
  Lab based algorithm: time until failure to maintain metabolic control (HbA1c level >= 7.0% or 53 mmol/mol)

SECONDARY OUTCOMES:
Time until a severe hypoglycemic episode | Through censoring or study completion, up to 765 day after cohort entry
  Claims based algorithm: time until a severe hypoglycemic episode
HbA1C change from baseline | Through censoring or study completion, up to 765 days after cohort entry
  Lab based algorithm: HbA1C change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT05099198/Prot_SAP_000.pdf